CLINICAL TRIAL: NCT06094218
Title: Development of a Treatment Prognosis Calculator for the Prevention of Suicide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jay Fournier, Associate Professor, Department of Psychiatry & Behavioral Health, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022H0245
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-01

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is a two phase, stepped-wedge design. In Phase I, all participants receive TAU. In Phase II, sites are randomized to receive training in BCBT. Prior to the training, participants receive TAU. Following the training, participants may receive BCBT.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): TAU may include (1) routine suicide risk screening and assessment; (2) safety planning with means restriction; and (3) the Collaborative Assessment and Management of Suicidality (CAMS), an evidence-based approach to managing and treating suicidal patients.
  Interventions: Behavioral: Treatment as usual (TAU)
- Brief Cognitive Behavioral Therapy (BCBT) (Experimental): BCBT consists of 12 outpatient individual psychotherapy sessions scheduled weekly or biweekly. The first session is 90 minutes and subsequent sessions are 60 minutes. BCBT is divided into three phases. In phase 1 (5 sessions), the therapist conducts a detailed assessment of the patient's most recent suicidal episode or suicide attempt, identifies patient-specific factors that contribute to and maintain suicidal behaviors, provides a cognitive-behavioral conceptualization, collaboratively develops a crisis response plan, and teaches basic emotion regulation skills. In phase 2 (5 sessions), the therapist teaches cognitive restructuring skills to build cognitive flexibility. In phase 3 (2 sessions), a relapse prevention task is conducted, and participants must demonstrate the ability to successfully complete this task in order to terminate the treatment. Additional sessions are conducted until participants demonstrate the ability to successfully complete this task.
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy (BCBT)

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy (BCBT) — BCBT was developed to provide patients with the skills they need to better manage the cognitive, emotional, physiological, and behavioral components of acute suicidal crises.
  Arms: Brief Cognitive Behavioral Therapy (BCBT)
Behavioral: Treatment as usual (TAU) — Behavioral health treatment as it is typically provided at the treatment site.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this interventional study is to develop and test a treatment prognosis calculator to identify which service members with suicidal ideation or behavior are likely to respond well to the current standard of care treatment and which should instead receive Brief Cognitive Behavioral Therapy (BCBT) as a first-line treatment.

The main aims of the study are:

* Aim 1: To develop a novel treatment prognostic calculator to predict response to treatment as usual (TAU) and identify treatment-seeking military personnel who are unlikely to respond adequately to TAU for the reduction of suicidal ideation.
* Aim 2: To evaluate the performance of the treatment prognosis calculator in a new sample of treatment-seeking military personnel and determine whether BCBT is more effective than TAU for those patients who are predicted not to respond adequately to TAU.

Participants will receive mental health treatment as it is typically administered by their mental healthcare treatment team. Members of their mental healthcare treatment team may receive intensive training in BCBT. After their provider has received this training, they may use this treatment as part of standard of care treatment. The timing of this training will be determined randomly. Participants will complete self-report assessments at the beginning of the study (baseline) as well as 3, 6, 9 and 12 months after their participant begins. These assessments will include questions about feelings, thoughts, moods, impulses, substance use, and behavior.

ELIGIBILITY:
Inclusion Criteria:

1. female and male active duty service members;
2. => 18 years old;
3. engaged in mental health treatment at one of the sites at study enrollment;
4. score >0 on the Columbia Suicide Severity Rating Scale (CSSRS) Screener-Recent, or indicated suicidal ideation on questions 4 or 5 of the Scale for Suicidal Ideation, indicating suicidal ideation within the last month;
5. able to understand and speak English;
6. able to provide consent.

Exclusion Criteria:

(1) participants with a psychiatric or medical condition that prevents them from providing informed consent or from participating in the treatments (e.g., psychosis, mania, acute intoxication).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | 6 Months
  Assess severity of suicidal ideation at 6 months with the Scale for Suicide Ideation (SSI)

SECONDARY OUTCOMES:
Suicide Attempts | 12 Months
  Suicide attempts will be assessed with the Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R)
Depression | 12 Months
  Depression will be assessed with the PROMIS-Depression Computer Adaptive Test (CAT)
Hopelessness | 12 Months
  Hopelessness will be assessed with the abbreviated Beck Hopelessness Scale (BHS)

CONTACTS AND LOCATIONS:
Locations (1):
- Harding Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No